CLINICAL TRIAL: NCT00217737
Title: A Randomized Phase III Study Comparing 5-FU, Leucovorin and Oxaliplatin Versus 5-FU, Leucovorin, Oxaliplatin and Bevacizumab in Patients With Stage II Colon Cancer at High Risk for Recurrence to Determine Prospectively the Prognostic Value of Molecular Markers
Brief Title: Oxaliplatin, Leucovorin, and Fluorouracil With or Without Bevacizumab in Treating Patients Who Have Undergone Surgery for Stage II Colon Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00562; NCI-2009-00562 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 05-198; CDR0000443410; E5202; ECOG-E5202; E5202 (Other: ECOG-ACRIN Cancer Research Group); E5202 (Other: CTEP); U10CA021115 (NIH); U10CA180820 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2025-07-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Colon Adenocarcinoma; Stage IIA Colon Cancer AJCC v7; Stage IIB Colon Cancer AJCC v7; Stage IIC Colon Cancer AJCC v7
MeSH Terms: conditions — Colonic Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Fluorouracil; dehydroftorafur; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (5-FU, leucovorin, oxaliplatin) (Active Comparator): Patients receive oxaliplatin IV over 2 hours and leucovorin IV over 2 hours on day 1. Patients also receive fluorouracil IV continuously over 46 hours beginning on day 1. Treatment repeats every 2 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- Arm B (5-FU, leucovorin, oxaliplatin, bevacizumab) (Experimental): Patients receive oxaliplatin, leucovorin, and fluorouracil as in Arm A and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 2 weeks for 12 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab alone for 12 additional courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- Arm C (observation) (No Intervention): Patients undergo observation.

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm B (5-FU, leucovorin, oxaliplatin, bevacizumab)
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm A (5-FU, leucovorin, oxaliplatin); Arm B (5-FU, leucovorin, oxaliplatin, bevacizumab)
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
  Arms: Arm A (5-FU, leucovorin, oxaliplatin); Arm B (5-FU, leucovorin, oxaliplatin, bevacizumab)
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
  Arms: Arm A (5-FU, leucovorin, oxaliplatin); Arm B (5-FU, leucovorin, oxaliplatin, bevacizumab)

SUMMARY:
This randomized phase III trial studies oxaliplatin, leucovorin, fluorouracil, and bevacizumab to see how well they work compared to oxaliplatin, leucovorin, and fluorouracil in treating patients who have undergone surgery for stage II colon cancer. Drugs used in chemotherapy, such as oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. It is not yet known whether giving combination chemotherapy together with bevacizumab is more effective than combination chemotherapy alone in treating colon cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate an improvement in 3-year disease-free survival for high-risk stage II colon cancer patients randomly assigned to 5-FU (fluorouracil), leucovorin, oxaliplatin versus 5-FU, leucovorin, oxaliplatin and bevacizumab.

SECONDARY OBJECTIVES:

I. To compare overall survival between the regimens. II. To further define the toxicity profiles of the regimens. III. To prospectively determine the impact of tumor biological characteristics on the survival of patients with stage II colon cancer.

IV. To assess the association between oxaliplatin exposure, allelic variants in candidate genes, and neurotoxicity. (Pharmacogenetic ancillary objective)

OUTLINE: Patients with high-risk disease are randomized to 1 of 2 treatment arms (Arms A and B). Patients with low-risk disease are assigned to Arm C.

ARM A: Patients receive oxaliplatin intravenously (IV) over 2 hours and leucovorin IV over 2 hours on day 1. Patients also receive fluorouracil IV continuously over 46 hours beginning on day 1. Treatment repeats every 2 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive oxaliplatin, leucovorin, and fluorouracil as in Arm A and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 2 weeks for 12 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab alone for 12 additional courses in the absence of disease progression or unacceptable toxicity.

ARM C: Patients undergo observation.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then every 12 months for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1: INITIAL REGISTRATION
* The distal extent of the tumor must be >= 12 cm from the anal verge on endoscopy; if this distance was not confirmed on endoscopy pre-operatively, then the distal extent of the tumor must be >= 12 cm from the anal verge as determined by surgical examination; colonoscopy should be performed postoperatively for those unable to have a preoperative colonoscopy to guarantee there are no synchronous lesions
* Patients must have paraffin-embedded tumor specimen available for evaluation of microsatellite instability and loss of heterozygosity at 18q, to determine high risk versus low risk

  * High-risk patients will be randomized to treatment Arms A or B
  * Low-risk patients will be registered to Arm C for observation

    * NOTE: Every effort should be made to submit blocks (tumor and normal mucosa) to the Principal Coordinates Analysis (PCO) immediately; blocks CANNOT be accepted after day 50 (post surgery) in order to allow for molecular assessment
    * Specific laboratory requirements for Step 2 must be obtained within 2 weeks prior to Step 2 randomization
* Patients must not have synchronous tumors
* Patients must not have appendiceal tumors
* Patients must not have a history of inflammatory bowel disease (IBD)
* Patients with hereditary non-polyposis colorectal cancer (HNPCC) are eligible
* Patients must have no history of isolated, distant, or non-contiguous intra-abdominal metastases, even if restricted
* Patients must have histologically confirmed adenocarcinoma of the colon that meets the criteria below:

  * Stage II adenocarcinoma (pT3/pT4a/pT4b pN0 M0 according to the definitions of the American Joint Committee on Cancer, 7th Edition, 2010): the tumor invades through the muscularis propria into pericolic tissues (pT3), penetrates to the surface of the visceral peritoneum (pT4a), or directly invades other organs or structures (pT4b); patients with mesenteric tumor deposits or satellites without identifiable residual lymph node in the absence of lymph node involvement are now designated pN1c, rather than pT3; patients with such tumor deposits are not eligible for E5202; patients must have had a complete resection (R0 resection)
* Patients must have >= 8 lymph nodes evaluated and reported
* Patients must not have presented with clinical complete obstruction or perforation of the bowel
* Patients must not have had any systemic or radiation therapy initiated for this malignancy
* Patients must not have a previous or concurrent malignancy; exceptions are made for patients who meet any of the following conditions:

  * Non-melanoma skin cancer, in situ cervical cancer, or breast cancer in situ
  * Prior malignancy completely excised or removed and patient has been continuously disease free for > 5 years
  * Patients with completely excised or removed breast cancer and disease free > 5 years, regardless of the continuation of hormonal therapy
  * Patients with previous radiation therapy (RT) to the pelvic region will be ineligible
* Patients must be ≥ 18 years old
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* STEP 2: RANDOMIZATION (HIGH RISK PATIENTS - ARMS A AND B ONLY)
* Within 2 weeks prior to randomization, postoperative absolute granulocyte count (AGC) must be >= 1500/mm^3 (or < 1500/mm^3, if in the opinion of the investigator, this represents an ethnic or racial variation of normal)
* Within 2 weeks prior to randomization, the postoperative platelet count must be >= 100,000/mm^3
* Within 2 weeks prior to randomization, there must be postoperative evidence of adequate hepatic function; bilirubin must be =< upper limit of normal (ULN) unless the patient has a chronic grade 1 bilirubin elevation due to Gilbert's disease or similar syndrome due to slow conjugation of bilirubin
* Within 2 weeks prior to randomization, there must be postoperative evidence of adequate hepatic function; alkaline phosphatase must be < 2.5 x ULN
* Within 2 weeks prior to randomization, there must be postoperative evidence of adequate hepatic function; aspartate transaminase (AST) must be < 1.5 x ULN
* Within 2 weeks prior to randomization, there must be postoperative evidence of adequate renal function; serum creatinine =< 1.5 x ULN
* Within 2 weeks prior to randomization, there must be postoperative evidence of adequate renal function; urine protein/creatinine (UPC) ratio of < 1.0; patients with a UPC ratio >= 1.0 must undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate < 1 gm of protein in order to participate
* Patients with any significant bleeding that is not related to the primary colon tumor within 6 months prior to study entry are not eligible
* Patients with gastroduodenal ulcer(s) determined to be active by endoscopy are not eligible
* Patients with a history of hypertension must measure < 150/90 mmHg and be on a stable regimen of anti-hypertensive therapy
* Patients must not have a serious or non-healing wound, skin ulcers or bone fracture
* Patients experiencing clinically significant peripheral neuropathy at the time of step 2 randomization (defined in the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events version 4.0 [CTCAE 4.0] as grade 2 or greater neurosensory or neuromotor toxicity) are not eligible
* Patients must not have had invasive procedures, defined as follows:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to randomization
  * Core biopsy or other minor procedure, excluding placement of a vascular access device, within 7 days prior to randomization
  * Or anticipate the need for major surgical procedure(s) during the course of the study
* Patients must begin adjuvant treatment no less than 28 days and no more than 60 days from surgery
* Eligible patients of reproductive potential (both sexes) must agree to use an accepted and effective method of contraceptive during study therapy and for at least 3 months after the completion of bevacizumab; women must not be pregnant or breast-feeding because the study drugs administered may cause harm to an unborn fetus or breastfeeding child; all females of childbearing potential must have a serum pregnancy test to rule out pregnancy within 2 weeks prior to step 2 randomization
* Patients with prothrombin time (PT) (international normalized ratio [INR]) > 1.5 are not eligible, unless the patient is on full-dose anticoagulants; if so, the following criteria must be met for enrollment:

  * The subject must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin or on a stable dose of low molecular weight heparin
  * The subject must not have active bleeding or a pathological condition that is associated with a high risk of bleeding
* Patients with non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude any of the study therapy drugs are not eligible; specifically excluded are the following conditions:

  * New York Heart Association (NYHA) class III or IV congestive heart failure
  * Current symptomatic arrhythmia
  * Any non-malignant systemic disease
* Patients with a history of transient ischemic attack (TIA) or cerebrovascular accident (CVA) are not eligible
* Patients with a history of the following within twelve months of study entry are not eligible:

  * Arterial thromboembolic events
  * Unstable angina
  * Myocardial infarction
* Patients with symptomatic peripheral vascular disease are not eligible
* Patients with psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude them from meeting the study requirements are not eligible
* Patients must not have a known allergy to platinum compounds
* STEP 2: REGISTRATION (LOW-RISK PATIENTS - ARM C)
* Patients determined to be low risk are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2431 (Actual)
Dates: Start 2005-09-06 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2026-04-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Al B Benson, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (931):
- United States (913):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Providence Hospital, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - John Muir Medical Center-Concord, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Saint Jude Medical Center, Fullerton, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Saint Rose Hospital, Hayward, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Loma Linda Healthcare System, Loma Linda, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Providence Holy Cross Medical Center, Mission Hills, California
  - Memorial Medical Center, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Wilma Chan Highland Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - San Diego VA Medical Center, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Northbay Cancer Center, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Danbury Hospital, Danbury, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Broward Health North, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Cancer Centers of Central Florida PA, Leesburg, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Portneuf Medical Center, Pocatello, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - LaGrange Oncology Associates, Geneva, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Vigliotti, Antonio, P.G. M.D. (UIA Investigator), Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Franciscan St. James Health-Olympia Fields Campus, Olympia Fields, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Midwest Cancer Research Group Incorporated, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - MercyOne Genesis Davenport Cancer Center, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - HaysMed, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Our Lady Bellefonte Hospital, Ashland, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - DeSoto Regional Health System, Mansfield, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Saint Mary's Regional Medical Center, Lewiston, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - York Hospital, York Village, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Meritus Medical Center, Hagerstown, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Commonwealth Hematology Oncology PC-Concord, Concord, Massachusetts
  - Dana Farber Community Cancer Care-Haverhill, Haverhill, Massachusetts
  - Saints Memorial Medical Center, Lowell, Massachusetts
  - Lawrence Memorial, Medford, Massachusetts
  - Dana Farber-Merrimack Valley, Methuen, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Norwood Hospital, Norwood, Massachusetts
  - Dana Farber Community Cancer Care-Quincy, Quincy, Massachusetts
  - Dana Farber Community Cancer Care-Stoneham, Stoneham, Massachusetts
  - Morton Hospital and Medical Center, Taunton, Massachusetts
  - Dana Farber Community Cancer Care-Weymouth, Weymouth, Massachusetts
  - Commonwealth Hematology Oncology PC-Worcester, Worcester, Massachusetts
  - Reliant Medical Group Inc, Worcester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Lapeer Regional Hospital, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Hematology and Oncology Clinic, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - Veterans Administration, Columbia, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Freeman Health System, Joplin, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Internal Medicine of Bozeman, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Cancer Alliance of Nebraska, Omaha, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson-Tahoe Specialty Medical Center, Carson City, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Nevada Cancer Institute-Summerlin Campus, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Ocean University Medical Center, Brick, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - John F Kennedy Medical Center, Edison, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Mountainside Hospital, Montclair, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Saint Luke's Hospital-Warren Campus, Phillipsburg, New Jersey
  - AtlantiCare Regional Medical Center -Main Campus, Pomona, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Saint Francis Medical Center, Trenton, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Veteran Affairs New York Harbor Healthcare System-Brooklyn Campus, Brooklyn, New York
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Nyack Hospital, Nyack, New York
  - Rochester General Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Syracuse Veterans Administration Medical Center, Syracuse, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Lenoir Memorial Hospital, Kinston, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Person Memorial Hospital, Roxboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Cole, Sharon, K. M.D. (UIA Investigator), Kenton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Stark, Michael, Edward. M.D. (UIA Investigator), Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Saint John Medical Center, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, DuBois, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Temple Health - Chestnut Hill Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Hematology and Oncology Associates of Rhode Island Inc, Cranston, Rhode Island
  - Roger Williams Medical Center, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Jones Clinic, Germantown, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Tennessee Cancer Specialists-Dowell Springs, Knoxville, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - East Tennessee Baptist Hospital-Mercy Health Partners, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology-Austin North, Austin, Texas
  - Texas Oncology Seton Northwest, Austin, Texas
  - Texas Oncology-Cedar Park, Cedar Park, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Oncology- San Marcos, San Marcos, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Mount Ascutney Hospital and Health Center, Windsor, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - VA Puget Sound Health Care System, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Providence Holy Family Hospital, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Marshall University Medical Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Aurora Cancer Care-Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - UW Health Oncology-One South Park, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic - Slinger, Slinger, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (12):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Health Sciences North, Greater Sudbury, Ontario
  - London Regional Cancer Program, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - PEI Cancer Treatment Centre-Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Puerto Rico (4):
  - Andres Grillasca Hospital, Ponce
  - San Juan Community Oncology Group, San Juan
  - San Juan Veterans Affairs Medical Center, San Juan
  - San Juan City Hospital, San Juan
- University Of Pretoria, Pretoria, South Africa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on August 4th, 2005 and was closed to accrual on February 11th, 2011. A total of 2,431 patients were enrolled.
Groups:
- Arm A (5-FU, Leucovorin, Oxaliplatin): Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1. Patients also receive fluorouracil IV continuously over 46 hours beginning on day 1. Treatment repeats every 2 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.
- Arm B (5-FU, Leucovorin, Oxaliplatin, Bevacizumab): Patients receive oxaliplatin, leucovorin calcium, and fluorouracil as in Arm A and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 2 weeks for 12 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab alone for 12 additional courses in the absence of disease progression or unacceptable toxicity.
- No Randomization/Registration at Step 2: Patients whose risk assessment information was unavailable or who did not registered to Step 2 are included in this group.
Period: Step 1 Registration (Risk Assessment)
Arm/Group | Arm A (5-FU, Leucovorin, Oxaliplatin) | Arm B (5-FU, Leucovorin, Oxaliplatin, Bevacizumab) | Arm C (Observation) | No Randomization/Registration at Step 2
Started | 460 | 458 | 1013 | 500
Completed | 460 | 458 | 1013 | 0
Not Completed | 0 | 0 | 0 | 500
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 252
Not completed — No tumor block assessments | 0 | 0 | 0 | 83
Not completed — Ineligible | 0 | 0 | 0 | 68
Not completed — Uninformative tumor block | 0 | 0 | 0 | 18
Not completed — Physician Decision | 0 | 0 | 0 | 16
Not completed — Study suspension/closure before treatment | 0 | 0 | 0 | 16
Not completed — Staff/site error | 0 | 0 | 0 | 9
Not completed — Unable to follow treatment schedule | 0 | 0 | 0 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 6
Not completed — Insurance issues | 0 | 0 | 0 | 4
Not completed — Non-compliance | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Disease progression | 0 | 0 | 0 | 1
Not completed — Inadequate supply of Leucovorin | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 12
Not completed — Registration error | 0 | 0 | 0 | 1
Period: Step 2 Randomization/Registration
Arm/Group | Arm A (5-FU, Leucovorin, Oxaliplatin) | Arm B (5-FU, Leucovorin, Oxaliplatin, Bevacizumab) | Arm C (Observation) | No Randomization/Registration at Step 2
Started | 460 | 458 | 1013 | 0
Eligible Patients | 424 | 435 | 998 | 0
Received Treatment | 429 | 410 | 0 | 0
Received Treatment and Toxicity Data Available | 428 | 410 | 0 | 0
Included in the Analysis of Impact of Tumor Biological Characteristics on Survival | 326 | 324 | 718 | 0
Completed | 304 | 143 | 1013 | 0
Not Completed | 156 | 315 | 0 | 0
Not completed — Adverse Event | 59 | 98 | 0 | 0
Not completed — Withdrawal by Subject | 53 | 105 | 0 | 0
Not completed — Study suspension | 0 | 45 | 0 | 0
Not completed — Complicating disease | 5 | 5 | 0 | 0
Not completed — Death | 2 | 3 | 0 | 0
Not completed — Non-compliant | 2 | 4 | 0 | 0
Not completed — Physician Decision | 2 | 2 | 0 | 0
Not completed — Alternative therapy | 0 | 1 | 0 | 0
Not completed — Extraordinary Medical Circumstances | 0 | 1 | 0 | 0
Not completed — Found to be Ineligible After Treatment | 0 | 1 | 0 | 0
Not completed — Incorrect Cancer Stage | 1 | 0 | 0 | 0
Not completed — Never started protocol therapy | 31 | 48 | 0 | 0
Not completed — Other | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients registered to Step 2 are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (5-FU, Leucovorin, Oxaliplatin) | Arm B (5-FU, Leucovorin, Oxaliplatin, Bevacizumab) | Arm C (Observation) | Total
Number analyzed (Participants) | 460 | 458 | 1013 | 1931
Age, Continuous [Median (Full Range); unit: years] | 59 [26 to 87] | 59 [25 to 85] | 60 [19 to 90] | 60 [19 to 90]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient with unknown sex was excluded from the analysis of distribution of sex.
  Participants
    number analyzed (Participants) | 459 | 458 | 1013 | 1930
    Female | 235 | 232 | 496 | 963
    Male | 224 | 226 | 517 | 967
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 32 | 88 | 149
  Not Hispanic or Latino | 401 | 390 | 868 | 1659
  Unknown or Not Reported | 30 | 36 | 57 | 123
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 17 | 14 | 32 | 63
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 49 | 55 | 85 | 189
  White | 385 | 372 | 882 | 1639
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 6 | 15 | 14 | 35

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival Rate at 5 Years
Description: Disease-free survival (DFS) is defined as the time from randomization to the earlier of disease recurrence, new invasive primary cancer, or death from any cause. The Kaplan-Meier estimates were used to characterize the 5-year DFS rates.
Time Frame: Assessed every 3 months for patients within 2 years of step 2 randomization, every 6 months during 3-5 years from step 2 randomization, and then every 12 months until 10 years from step 2 randomization
Population: Eligible patients who were registered or randomized at Step 2 were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A (5-FU, Leucovorin, Oxaliplatin) | Arm B (5-FU, Leucovorin, Oxaliplatin, Bevacizumab) | Arm C (Observation)
Number analyzed (Participants) | 424 | 435 | 998
Proportion of participants | 0.805 [0.766 to 0.846] | 0.833 [0.796 to 0.871] | 0.816 [0.791 to 0.842]
Statistical Analysis 1: Comparison: Arm A (5-FU, Leucovorin, Oxaliplatin) vs Arm B (5-FU, Leucovorin, Oxaliplatin, Bevacizumab); Test type: Superiority; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.63 to 1.11] — Hazard ratio: Arm B/Arm A

2. Secondary Outcome: Overall Survival Rate at 5 Years
Description: Overall survival (OS) is defined as the time from randomization to death from any cause. OS is censored at the date of last contact for patients still alive. The Kaplan-Meier estimates were used to characterize the 5-year OS rates.
Time Frame: as for outcome 1
Population: Eligible patients who were registered or randomized at Step 2 were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A (5-FU, Leucovorin, Oxaliplatin) | Arm B (5-FU, Leucovorin, Oxaliplatin, Bevacizumab) | Arm C (Observation)
Number analyzed (Participants) | 424 | 435 | 998
Proportion of participants | 0.918 [0.891 to 0.946] | 0.921 [0.895 to 0.948] | 0.926 [0.909 to 0.943]

3. Secondary Outcome: The Impact of Tumor Biological Characteristics on Overall Survival
Description: Overall survival (OS) is defined as the time from randomization to death from any cause. OS is censored at the date of last contact for patients still alive. The following patient/tumor characteristics were associated with overall survival:
  * ECOG Performance Status (0, 1, or 2)
  * Age
  * Sex (male, female)
  * Primary tumor site (right-side colon, transverse colon, left-side colon, or other)
  * Number of regional lymph nodes
  Hazard ratios with adjustment for other covariates are reported with OS as the outcome variable.
Time Frame: Assessed at baseline, every 3 months for patients within 2 years of step 2 randomization, every 6 months during 3-5 years from step 2 randomization, and then every 12 months until 10 years from step 2 randomization
Population: Eligible patients who had advanced to step 2 (Arms A, B and C) and had complete data on patient/tumor characteristics are included.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Groups:
- Tumor Biological Characteristics and Overall Survival Analysis: Eligible patients who had advanced to step 2 (Arms A, B and C) and had complete data on patient/tumor characteristics are included.
Arm/Group | Tumor Biological Characteristics and Overall Survival Analysis
Number analyzed (Participants) | 1368
hazard ratio
  Hazard ratio: ECOG performance status of 1 (vs. 0) | 1.67 [1.24 to 2.25]
  Hazard ratio: ECOG performance status of 2 (vs. 0) | 3.39 [1.36 to 8.44]
  Hazard ratio: Age | 1.05 [1.04 to 1.07]
  Hazard ratio: Sex of male (vs. female) | 1.71 [1.27 to 2.28]
  Hazard ratio: Primary site of transverse colon (vs. Right-side colon) | 0.81 [0.44 to 1.52]
  Hazard ratio: Primary site of left-side colon (vs. Right-side colon) | 1.13 [0.82 to 1.55]
  Hazard ratio: Primary site of other (vs. Right-side colon) | 2.68 [1.39 to 5.17]
  Hazard ratio: Number of lymph nodes | 0.98 [0.96 to 0.99]

4. Other Pre Specified Outcome: The Association Between Oxaliplatin Exposure, Allelic Variants in Candidate Genes, and Neurotoxicity
Description: The association between onset of neurotoxicity and oxaliplatin exposure will be assessed. The difference in neurotoxicity rates between patients with and without a given polymorphism will be evaluated.
Time Frame: Assessed at baseline, every 2 weeks while on treatment, up to 10 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 2 weeks while on treatment and for 30 days after the end of treatment, up to 10 years
Description: All patients received treatment at Step 2 and had adverse event data were included in the analysis of adverse events. Patients who underwent observation in Arm C did not receive any treatment, so no adverse event data were collected for these patients.
  All patients registered/randomized at Step 2 were included in the analysis of all-cause mortality.
Arm/Group | Arm A (5-FU, Leucovorin, Oxaliplatin) | Arm B (5-FU, Leucovorin, Oxaliplatin, Bevacizumab) | Arm C (Observation) | No Randomization/Registration at Step 2
All-Cause Mortality (participants affected / at risk) | 73/460 | 69/458 | 145/1013 | 61/500
Serious Adverse Events (participants affected / at risk) | 308/428 | 292/410 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 399/428 | 388/410 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (5-FU, Leucovorin, Oxaliplatin) (N=428) | Arm B (5-FU, Leucovorin, Oxaliplatin, Bevacizumab) (N=410) | Arm C (Observation) (N=0) | No Randomization/Registration at Step 2 (N=0)
Allergic reaction (Immune system disorders) | 12 | 7 | NA | NA
Hearing w/o audiogr not in monitor prg (Ear and labyrinth disorders) | 1 | 1 | NA | NA
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 0 | 2 | NA | NA
Anemia (Blood and lymphatic system disorders) | 3 | 1 | NA | NA
Leukocytes decreased (Investigations) | 42 | 29 | NA | NA
Lymphopenia (Investigations) | 3 | 3 | NA | NA
Neutrophils decreased (Investigations) | 178 | 138 | NA | NA
Platelets decreased (Investigations) | 18 | 3 | NA | NA
Arrhythmia-other (Cardiac disorders) | 0 | 2 | NA | NA
Cardiac-ischemia (Cardiac disorders) | 3 | 2 | NA | NA
Cardiac troponin I (cTnI) increased (Investigations) | 0 | 1 | NA | NA
Hypertension (Vascular disorders) | 1 | 36 | NA | NA
Hypotension (Vascular disorders) | 4 | 2 | NA | NA
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 1 | NA | NA
Cardiomyopathy, restrictive (Cardiac disorders) | 0 | 1 | NA | NA
Valvular heart disease (Cardiac disorders) | 0 | 1 | NA | NA
Fatigue (General disorders) | 33 | 41 | NA | NA
Fever w/o neutropenia (General disorders) | 0 | 1 | NA | NA
Insomnia (Psychiatric disorders) | 3 | 0 | NA | NA
Rigors/chills (General disorders) | 1 | 1 | NA | NA
Weight gain (Investigations) | 0 | 1 | NA | NA
INR increased (Investigations) | 2 | 3 | NA | NA
Coagulation-other (Investigations) | 0 | 2 | NA | NA
Injection site reaction (General disorders) | 1 | 0 | NA | NA
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 5 | NA | NA
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 7 | 16 | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Wound - non-infectious (Injury, poisoning and procedural complications) | 0 | 3 | NA | NA
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Death - multiorgan failure (General disorders) | 0 | 2 | NA | NA
Pancreatic glucose intolerance (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Anorexia (Metabolism and nutrition disorders) | 4 | 11 | NA | NA
Colitis (Gastrointestinal disorders) | 0 | 2 | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 1 | NA | NA
Dehydration (Metabolism and nutrition disorders) | 14 | 18 | NA | NA
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 47 | 55 | NA | NA
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 1 | NA | NA
Dysphagia (Gastrointestinal disorders) | 0 | 1 | NA | NA
Esophagitis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Fistula, Rectum (Gastrointestinal disorders) | 0 | 1 | NA | NA
Gastritis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | NA | NA
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | NA | NA
Ileus (Gastrointestinal disorders) | 4 | 3 | NA | NA
Leak, incl. anastomotic, large bowel (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 9 | 5 | NA | NA
Muco/stomatitis by exam, pharynx (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | NA | NA
Muco/stomatitis (symptom) anus (Gastrointestinal disorders) | 0 | 1 | NA | NA
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 6 | 7 | NA | NA
Muco/stomatitis (symptom) pharynx (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | NA | NA
Nausea (Gastrointestinal disorders) | 17 | 22 | NA | NA
Necrosis, gallbladder (Hepatobiliary disorders) | 1 | 0 | NA | NA
Obstruction, small bowel NOS (Gastrointestinal disorders) | 0 | 1 | NA | NA
Perforation, appendix (Infections and infestations) | 0 | 1 | NA | NA
Perforation, ileum (Gastrointestinal disorders) | 0 | 1 | NA | NA
Perforation, small bowel NOS (Gastrointestinal disorders) | 1 | 1 | NA | NA
Stenosis (incl anastomotic) colon (Gastrointestinal disorders) | 0 | 1 | NA | NA
Typhlitis (Gastrointestinal disorders) | 0 | 2 | NA | NA
Vomiting (Gastrointestinal disorders) | 11 | 11 | NA | NA
GI-other (Gastrointestinal disorders) | 0 | 1 | NA | NA
CNS, hemorrhage (Nervous system disorders) | 0 | 1 | NA | NA
Colon, hemorrhage (Gastrointestinal disorders) | 0 | 1 | NA | NA
Lower GI, hemorrhage NOS (Gastrointestinal disorders) | 0 | 1 | NA | NA
Upper GI, hemorrhage NOS (Gastrointestinal disorders) | 0 | 1 | NA | NA
Urinary hemorrhage NOS (Renal and urinary disorders) | 0 | 1 | NA | NA
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Surgical hemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | NA | NA
Liver dysfunction/failure (Hepatobiliary disorders) | 0 | 1 | NA | NA
Colitis, infectious (e.g. C.diff) (Infections and infestations) | 1 | 0 | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 0 | NA | NA
Infection w/ gr3-4 neut, catheter relate (Infections and infestations) | 1 | 0 | NA | NA
Infection w/ gr3-4 neut, ileum (Infections and infestations) | 0 | 1 | NA | NA
Infection w/ gr3-4 neut, lung (Infections and infestations) | 1 | 0 | NA | NA
Infection Gr0-2 neut, abdomen (Infections and infestations) | 0 | 1 | NA | NA
Infection Gr0-2 neut, appendix (Infections and infestations) | 0 | 1 | NA | NA
Infection Gr0-2 neut, bronchus (Infections and infestations) | 0 | 1 | NA | NA
Infection Gr0-2 neut, catheter (Infections and infestations) | 2 | 3 | NA | NA
Infection Gr0-2 neut, colon (Infections and infestations) | 1 | 1 | NA | NA
Infection Gr0-2 neut, gallbladder (Infections and infestations) | 1 | 0 | NA | NA
Infection Gr0-2 neut, lung (Infections and infestations) | 2 | 1 | NA | NA
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 0 | 1 | NA | NA
Infection Gr0-2 neut, peritoneal (Infections and infestations) | 0 | 1 | NA | NA
Infection Gr0-2 neut, skin (Infections and infestations) | 1 | 0 | NA | NA
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 0 | 1 | NA | NA
Opportunistic infection lymphopenia>=gr1 (Infections and infestations) | 1 | 0 | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1 | NA | NA
Alanine aminotransferase increased (Investigations) | 2 | 4 | NA | NA
Serum amylase increased (Investigations) | 0 | 1 | NA | NA
Aspartate aminotransferase increased (Investigations) | 3 | 4 | NA | NA
Blood bilirubin increased (Investigations) | 1 | 0 | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2 | NA | NA
Hypercholesterolemia (Investigations) | 0 | 1 | NA | NA
Creatinine increased (Investigations) | 1 | 3 | NA | NA
GGT increased (Investigations) | 1 | 0 | NA | NA
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 4 | NA | NA
Lipase increased (Investigations) | 0 | 1 | NA | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | NA | NA
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2 | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 14 | 13 | NA | NA
Proteinuria (Renal and urinary disorders) | 0 | 5 | NA | NA
Hyponatremia (Metabolism and nutrition disorders) | 3 | 7 | NA | NA
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Metabolic/Laboratory-other (Investigations) | 0 | 1 | NA | NA
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Nonneuropathic upper extr muscle weak (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Soft tissue necrosis, head (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 0 | NA | NA
Dizziness (Nervous system disorders) | 0 | 4 | NA | NA
Laryngeal nerve dysfunction (Nervous system disorders) | 1 | 0 | NA | NA
Mental status (Nervous system disorders) | 0 | 1 | NA | NA
Depression (Psychiatric disorders) | 2 | 0 | NA | NA
Neuropathy CN V jaw / face-sensory (Nervous system disorders) | 1 | 0 | NA | NA
Neuropathy-motor (Nervous system disorders) | 3 | 2 | NA | NA
Neuropathy-sensory (Nervous system disorders) | 80 | 78 | NA | NA
Seizure (Nervous system disorders) | 0 | 1 | NA | NA
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | NA | NA
Syncope (Nervous system disorders) | 1 | 6 | NA | NA
Tremor (Nervous system disorders) | 0 | 1 | NA | NA
Neurologic-other (Nervous system disorders) | 6 | 5 | NA | NA
Vision-flashing lights/floaters (Eye disorders) | 1 | 0 | NA | NA
Ocular-other (Eye disorders) | 1 | 0 | NA | NA
Abdomen, pain (Gastrointestinal disorders) | 7 | 12 | NA | NA
Back, pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | NA | NA
Bone, pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Buttock, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Cardiac/heart, pain (Cardiac disorders) | 0 | 1 | NA | NA
Chest/thoracic pain NOS (General disorders) | 2 | 1 | NA | NA
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Gallbladder, pain (Hepatobiliary disorders) | 1 | 0 | NA | NA
Head/headache (Nervous system disorders) | 5 | 4 | NA | NA
Joint, pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | NA | NA
Muscle, pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | NA | NA
Neck, pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Oral cavity, pain (Gastrointestinal disorders) | 1 | 0 | NA | NA
Pain NOS (General disorders) | 1 | 0 | NA | NA
Pleura, pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pain-other (General disorders) | 0 | 1 | NA | NA
(ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | NA | NA
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | NA | NA
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | NA | NA
Renal failure (Renal and urinary disorders) | 1 | 2 | NA | NA
Cytokine release syndrome (Immune system disorders) | 2 | 0 | NA | NA
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 7 | 11 | NA | NA
Thrombosis/thrombus/embolism (Vascular disorders) | 9 | 19 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (5-FU, Leucovorin, Oxaliplatin) (N=428) | Arm B (5-FU, Leucovorin, Oxaliplatin, Bevacizumab) (N=410) | Arm C (Observation) (N=0) | No Randomization/Registration at Step 2 (N=0)
Anemia (Blood and lymphatic system disorders) | 235 | 205 | NA | NA
Leukocytes decreased (Investigations) | 222 | 174 | NA | NA
Neutrophils decreased (Investigations) | 184 | 156 | NA | NA
Platelets decreased (Investigations) | 227 | 152 | NA | NA
Hypertension (Vascular disorders) | 12 | 111 | NA | NA
Fatigue (General disorders) | 294 | 278 | NA | NA
Insomnia (Psychiatric disorders) | 36 | 30 | NA | NA
Weight loss (Investigations) | 19 | 33 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 102 | 85 | NA | NA
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 13 | 21 | NA | NA
Nail changes (Skin and subcutaneous tissue disorders) | 11 | 22 | NA | NA
Rash/desquamation (Skin and subcutaneous tissue disorders) | 45 | 50 | NA | NA
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 62 | 56 | NA | NA
Anorexia (Metabolism and nutrition disorders) | 116 | 125 | NA | NA
Constipation (Gastrointestinal disorders) | 85 | 90 | NA | NA
Dehydration (Metabolism and nutrition disorders) | 23 | 35 | NA | NA
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 216 | 213 | NA | NA
Dyspepsia (Gastrointestinal disorders) | 22 | 33 | NA | NA
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 98 | 93 | NA | NA
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 69 | 75 | NA | NA
Nausea (Gastrointestinal disorders) | 240 | 233 | NA | NA
Taste disturbance (Nervous system disorders) | 67 | 62 | NA | NA
Vomiting (Gastrointestinal disorders) | 88 | 104 | NA | NA
Rectum, hemorrhage (Gastrointestinal disorders) | 4 | 27 | NA | NA
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 31 | 107 | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 33 | 29 | NA | NA
Alkaline phosphatase increased (Investigations) | 57 | 32 | NA | NA
Alanine aminotransferase increased (Investigations) | 68 | 48 | NA | NA
Aspartate aminotransferase increased (Investigations) | 88 | 62 | NA | NA
Blood bilirubin increased (Investigations) | 22 | 12 | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 28 | 32 | NA | NA
Creatinine increased (Investigations) | 7 | 23 | NA | NA
Hyperglycemia (Metabolism and nutrition disorders) | 43 | 48 | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 36 | 43 | NA | NA
Proteinuria (Renal and urinary disorders) | 7 | 61 | NA | NA
Hyponatremia (Metabolism and nutrition disorders) | 20 | 28 | NA | NA
Dizziness (Nervous system disorders) | 26 | 29 | NA | NA
Neuropathy-sensory (Nervous system disorders) | 331 | 286 | NA | NA
Neurologic-other (Nervous system disorders) | 33 | 27 | NA | NA
Abdomen, pain (Gastrointestinal disorders) | 39 | 51 | NA | NA
Head/headache (Nervous system disorders) | 45 | 76 | NA | NA
Joint, pain (Musculoskeletal and connective tissue disorders) | 9 | 28 | NA | NA
Muscle, pain (Musculoskeletal and connective tissue disorders) | 37 | 46 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 26 | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 29 | 50 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-04-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT00217737/Prot_SAP_000.pdf
  • Informed Consent Form (2014-04-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT00217737/ICF_001.pdf